CLINICAL TRIAL: NCT02902237
Title: Phase I Study of tTF-NGR in Patients With Recurrent or Refractory Malignant Tumors and Lymphomas Beyond All Standard Treatments
Brief Title: tTF-NGR Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM12_0018; 2016-003042-85 (EudraCT Number)
Record Dates: First submitted 2016-09-05; First posted 2016-09-15 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2019-04

CONDITIONS: Malignant Solid Tumors; Lymphomas
Keywords: tTF-NGR; vascular targeting; CD13; aminopeptidase N; first-in-class phase I study
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: Single-arm, mono-center, open-label phase I trial with intraindividual dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tTF-NGR (Experimental): tTF-NGR will be given as 1-hour infusion via central venous access once daily for 5 days with a subsequent rest period of 2 weeks and following cycles with dose escalation of 0.5 mg/m2 upon judgement of tolerability and therapeutic activity. Starting dose will be 1 mg/m2/day. Dose-escalation is stopped before the maximum number of 8 escalation steps if tumor response, tumor progression or a Dose-Limiting Toxicity (DLT) is observed.
  Interventions: Biological: tTF-NGR

INTERVENTIONS:
Biological: tTF-NGR — tTF-NGR will be given as 1-hour infusion via central venous access once daily for 5 days with a subsequent rest period of 2 weeks and following cycles with dose escalation of 0.5 mg/m2 upon judgement of tolerability and therapeutic activity. Starting dose will be 1 mg/m2/day. Dose-escalation is stopped before the maximum number of 8 escalation steps if tumor response, tumor progression or a Dose-Limiting Toxicity (DLT) is observed.
  Other Names: truncated tissue factor (tTF)-NGR

SUMMARY:
In this phase I clinical trial cancer patients suffering from solid tumors or lymphomas, recurring after and/or refractory against standard treatment are treated intravenously (iv) with increasing doses of tTF-NGR(tTF= truncated tissue factor; NGR=Asn-Gly-Arg). The objectives of this trial are to evaluate the maximum tolerated dose (MTD) and the dose-limiting toxicity (DLT) of intravenously (iv) infused daily applications of tTF-NGR for 5 days every 3 weeks in patients with cancer, who had obtained all standard treatment known for their disease entity prior to entry on study. Further objectives are to determine the perfusion and vascular volume fraction of measurable tumor lesions versus normal reference tissue before and after tTF-NGR application by MRI as a biological surrogate parameter for biological activity of the investigational medicinal product (IMP), tTF-NGR, and to obtain pharmacokinetic data.

DETAILED DESCRIPTION:
PHASE I STUDY OF tTF-NGR IN PATIENTS WITH RECURRENT OR REFRACTORY MALIGNANT TUMORS OR LYMPHOMAS BEYOND ALL STANDARD TREATMENTS

Short Title: tTF-NGR Phase I Study Sponsor's Study Code: UKM12_0018

EudraCT-No.: 2016-003042-85 Sponsor: Universitätsklinikum Muenster Investigator: Prof. Dr. Christoph Schliemann

Indication: All solid tumors and lymphomas beyond standard therapy Study Design: Phase I Study Investigational Medicinal Product: tTF-NGR

Therapy: Phase I, open label, single arm, non-randomized prospective, monocenter study. tTF-NGR will be given as 1-hour infusion via central venous access once daily for 5 days with a subsequent rest period of 2 weeks and following cycles with dose escalation of 0.5 mg/m2 upon judgement of tolerability and therapeutic activity. Starting dose will be 1 mg/m2/day. Patients within the dose-escalation part will be treated in sequence and not in parallel. Individual patients can undergo a maximum of 8 dose-escalations. Dose-escalation is stopped before the maximum number of 8 escalation steps if tumor response, tumor progression or a Dose-Limiting Toxicity (DLT) is observed. In the case of stable disease (SD) and with good tolerability these patients can obtain further cycles without dose-escalation until tumor progression or Dose-Limiting Toxicity (DLT) and the next patient can start with dose-escalation cycles on the highest tolerable dose for the previous patient.

Objectives:

Primary Objective:

To evaluate the maximum tolerated dose (MTD) and the Dose-Limiting Toxicity (DLT) of intravenously (iv) infused daily applications of tTF-NGR for 5 days every 3 weeks in patients with relapsed or refractory cancer, who had obtained all standard treatment known for their disease entity prior to entry on study.

Secondary Objectives:

1. To determine the perfusion and vascular volume fraction of measurable tumor lesions versus normal reference tissue before and after tTF-NGR application as a biological surrogate parameter for biological activity of the IMP in the patients treated within the verification cohorts.
2. To obtain pharmacokinetic data of tTF-NGR.

Endpoints:

Primary Safety Endpoint: Maximum Tolerated Dose (MTD). MTD is the dose below the dose leading to reproducible episodes of Dose Limiting Toxicity (DLT) in at least 2/6 patients. DLT will be characterized by clinical, blood and serum monitoring at specified time points before and during study period.

Secondary Efficacy Endpoints:

1. Occurrence and frequency of inhibition of tumor blood flow as measured by contrast-enhanced Magnetic Resonance Imaging (MRI) in the patients treated in the verification cohorts.
2. Occurrence and frequency of tumor response defined as Complete Response (CR), Partial Response (PR), or Stabile Disease (SD) as defined by RECIST criteria.

Inclusion Criteria:

* age > 18 years
* histologically proven or cytologically confirmed solid malignant tumor or malignant lymphoma
* recurrent or refractory disease after standard therapy and with no known curative or survival-prolonging treatment options according to the judgement of the investigators
* life expectancy of at least 6 weeks according to the judgement of the investigators
* Karnofsky performance status >50
* measurable disease with at least one marker-lesion measurable in 2 dimensions by Vascular Volume-Fraction-MRI
* adequate bone marrow function with absolute neutrophil count > 1000/microliter and platelet count > 50/nl.
* normal global coagulation parameters (Quick, PTT, TZ, fibrinogen), no prophylactic anticoagulation
* adequate liver function (total bilirubin < 3x the upper normal limit (ULN), SGPT/SGOT < 3x ULN)
* adequate renal function (serum creatinine < 3x ULN)
* no history of coronary heart disease, stroke, transitory ischemic attacks, pulmonary embolism, or deep vein thrombosis
* time elapsed from previous therapy (including other IMPs) > 3 weeks with recovery from side effects
* exclusion of central nervous system (CNS) disease and CNS vascular abnormalities by MRI
* ability to understand and provide written informed consent
* written informed consent given
* for female patients with child-bearing potential exclusion of pregnancy by adequate testing within 48 hours prior to entry on study
* females of childbearing potential as well as fertile males must agree to use a highly effective form of contraception (Pearl Index < 1) during the study and for 120 days following the last dose of the IMP

Exclusion Criteria:

* clinically significant unrelated illness which in the judgement of the investigators could compromise the patient's ability to tolerate the IMP or be likely to interfere with the study procedures or results
* known hypersensitivity reactions to prior application of E. coli-derived material
* women with breast-feeding activity
* concomitant use of any other investigational agent (agent for which there is currently no approved indication from regulatory authorities)
* clinical application of any other drug with known antitumor activity
* prophylactic anticoagulation within the last 3 days

NOTE: Since this is a phase I study for end-stage cancer patients, patients who would be excluded from the protocol strictly for laboratory abnormalities only can be included at the Investigator's discretion. This will be documented as an exception to the criteria and will be signed and filed in the CRF and the Trial Master File.

Statistical Methods: Descriptive statistics are performed to characterize MTD (= dose level below DLT occurring in 2/6 patients) Financial Support: Deutsche Krebshilfe, grant 111004 Schedule Planned start date of the study (FPFV): 01.11.2016 Planned end date of recruitment (LPFV): 01.11.2017 Planned end date of the study (LPLV): 01.05.2018

Studied period (years): (date of first enrolment) 2017 03 29; (date of last completed) 2019 12 19

Study centre: Department of Medicine A (Hematology, Hemostaseology, Oncology) University Hospital Muenster, Germany Albert-Schweitzer-Campus 1 D-48149 Muenster, Germany

Methodology:

We have treated 17 patients with advanced cancer beyond standard therapies with tTF-NGR applied as a 1-hour infusion via central venous access for 5 consecutive days and rest periods of 2 weeks before the next cycle. The study allowed for intraindividual dose escalations from cycle to cycle and established MTD and DLT by verification cohorts of 6 patients. This was an investigator-initiated, monocenter, single-arm, open-label study.

Number of patients (planned and analysed):

The number of patients required to complete this study was determined by the occurrence of DLT. Eventually, 24 patients had to be screened and 17 of them treated and analyzed in order to evaluate the study.

ELIGIBILITY:
Inclusion criteria:

* age ≥ 18 years
* histologically proven or cytologically confirmed solid malignant tumor or malignant lymphoma
* recurrent or refractory disease after standard therapy and with no known curative or survival-prolonging treatment options according to the judgement of the investigators
* life expectancy of at least 6 weeks according to the judgement of the investigators
* Karnofsky performance status ≥ 50
* measurable disease with at least one marker-lesion measurable in 2 dimensions by Vascular Volume-Fraction-MRI and/or CEUS.
* adequate bone marrow function with absolute neutrophil count > 1000/microliter and platelet count > 50/nl
* normal global coagulation parameters (Quick, partial thromboplastin time (PTT), thrombin time (TZ), fibrinogen), no prophylactic anticoagulation
* ability to understand and provide written informed consent
* adequate liver function (total bilirubin < 3x the upper normal limit (ULN), serum glutamic pyruvic transaminase/serum glutamic-oxaloacetic transaminase (SGPT/SGOT) < 3x ULN)
* adequate renal function (serum creatinine < 3x ULN)
* no history of coronary heart disease, stroke, transitory ischemic attacks, pulmonary embolism, or deep vein thrombosis
* time elapsed from previous therapy (including other IMPs) ≥ 3 weeks with recovery from side effects
* exclusion of central nervous system (CNS) disease and CNS vascular abnormalities by MRI
* ability to understand and provide written informed consent
* written informed consent given
* for female patients with child-bearing potential exclusion of pregnancy by adequate testing within 48 hours prior to entry on study
* females of childbearing potential as well as fertile males must agree to use a highly effective form of contraception (Pearl Index < 1) during the study and for 120 days following the last dose of the IMP

Exclusion criteria:

* clinically significant unrelated illness which in the judgement of the investigators could compromise the patient's ability to tolerate the IMP or be likely to interfere with the study procedures or results
* known hypersensitivity reactions to prior application of E. coli-derived material
* women with breast-feeding activity
* concomitant use of any other investigational agent (agent for which there is currently no approved indication from regulatory authorities)
* clinical application of any other drug with known anti tumor activity
* prophylactic anticoagulation within the last 3 days

NOTE: Since this is a phase I study for end-stage cancer patients, patients who would be excluded from the protocol strictly for laboratory abnormalities only can be included at the Investigator's discretion. This will be documented as an exception to the criteria and will be signed and filed in the CRF and the Trial Master File.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schliemann, Prof., Principal Investigator — University Hospital of Muenster
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcome measures will be made available within 6 months of study completion
Supporting Information: Study Protocol, SAP
Time Frame: Data are shared as a publication, June 2020
Access Criteria: Access to CANCERS necessary
URL: https://www.mdpi.com/2072-6694/12/6/1488

REFERENCES:
- [Result] Schliemann C, Gerwing M, Heinzow H, Harrach S, Schwoppe C, Wildgruber M, Hansmeier AA, Angenendt L, Berdel AF, Stalmann U, Berning B, Kratz-Albers K, Middelberg-Bisping K, Wiebe S, Albring J, Wilms C, Hartmann W, Wardelmann E, Krahling T, Heindel W, Gerss J, Bormann E, Schmidt H, Lenz G, Kessler T, Mesters RM, Berdel WE. First-In-Class CD13-Targeted Tissue Factor tTF-NGR in Patients with Recurrent or Refractory Malignant Tumors: Results of a Phase I Dose-Escalation Study. Cancers (Basel). 2020 Jun 7;12(6):1488. doi: 10.3390/cancers12061488. PMID 32517329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited in the University Hospital Muenster on an out-patient basis.
Pre-assignment Details: 24 patients were screened, 6 were screening failures(1: fast disease progression, 1: retraction of consent; 3: fast disease progression, 1: new brain metastasis diagnosed in screening). One patient died from sepsis before treatment with tTF-NGR, 17 patients obtained at least 1 application of tTF-NGR and were evaluable for safety, toxicity ans efficacy.
Period: Overall Study
Arm/Group | tTF-NGR
Started | 17
Completed | 17 (STUDY INITIATION: 2017 03 29, 1st Patient In, STUDY COMPLETION: 2019 11 05, Date of Study End)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Seventeen patients with advanced solid tumors beyond standard treatment.
Groups:
- tTF-NGR: This was a single-arm, mono-center, open-label trial. tTF-NGR was given as a 1-hour infusion via central venous access once daily for 5 days with a subsequent rest period of 2 weeks to all 17 patients treated. 8 patients received 2 cycles, 1 patient received 3 cycles, and 8 patients received 1 cycle.
Arm/Group | tTF-NGR
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 17
Disease type [Count of Participants; unit: Participants]
  germ cell tumor | 3
  hepatocellular tumor | 2
  lung tumor | 2
  colorectal tumor | 4
  soft tissue sarcoma | 5
  thyroid tumor | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Dose-limiting Toxicity (DLT)
Description: DLT will be characterized by clinical, blood and serum monitoring at specified time points before and during study period. AE, SAE, and SUSAR reporting was according to CTCAE 4.0 and GCP guidelines.
Time Frame: Measures: daily during treatment, weekly during rest periods of 2 weeks, monthly after End of Therapy, up to 3 months.
Population: All 17 patients treated with tTF-NGR were analysed for safety and toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- tTF-NGR: All 17 patients obtaining at least 1 dose of tTF-NGR were analysed for MTD and DLT.
Arm/Group | tTF-NGR
Number analyzed (Participants) | 17
Participants
  MTD (3 mg/m^2 tTF-NGR/day x 5, q day 22) | 8
  DLT: isolated and reversible elevation of Troponin T hs (grade 3 CTCAE 4.0) | 5
  other patient, who obtained other doses than MTD without DLT | 4

2. Secondary Outcome: 1: Assessment of Anti-tumor Activity: MRI K-trans in [ 10^-3/Min] and/or CEUS in [Arbitrary Units]; 2: Pharmacokinetic Profile: AUC in [ng*h/mL]
Description: 1: Anti-tumor activity: Tumor blood flow was measured with MRI and/or CEUS; 2: Pharmacokinetic data of tTF-NGR: tTF-NGR blood levels were analyzed by TF-ELISA.
Time Frame: 1: Tumor blood flow: baseline, 5 h post-dose, at 5 d at each cycle of therapy and 6 months. 2: Pharmacokinetic measures: 0 h, 0.5 h, 1 h, 1.5 h, 3 h, 2.5 h, 3 h, 3.5 h, 4 h, 4.5 h, 5 h post-dose
Population: All 17 patients obtaining at least 1 dose of tTF-NGR were analysed for efficacy and were assayed for tTF-NGR pharmacokinetics.
Measure: Count of Participants; unit: Participants
Groups:
- tTF-NGR: All 17 patients obtaining at least 1 dose of tTF-NGR were analysed for safety and efficacy. All 17 patients were assayed for tTF-NGR pharmacokinetics.
Arm/Group | tTF-NGR
Number analyzed (Participants) | 17
Participants
  Anti-tumor activity: blood flow reduction: yes | 17
  Anti-tumor activity: blood flow reduction: no | 0
  Pharmacokinetic profile: AUC determined: yes | 17
  Pharmacokinetic profile: AUC determined: no | 0

ADVERSE EVENTS:
Time Frame: All adverse events including serious adverse events were monitored from the first study-related procedure (tTF-NGR application) ,daily during treatment, weekly during rest periods of 2 weeks, monthly from the end of treatment with tTF-NGR up to 3 months.
Description: AE, SAE, SUSAR were classified according to CTCAE 4.0 criteria and reports were generated according to GCP guidelines.
Groups:
- tTF-NGR Dose: 1,0 mg/m^2; tTF-NGR Dose: 1,5 mg/m^2; tTF-NGR Dose: 2,0 mg/m^2; tTF-NGR Dose: 2,5 mg/m^2; tTF-NGR Dose: 3,0 mg/m^2; tTF-NGR Dose: 4,0 mg/m^2; tTF-NGR Dose: 5,0 mg/m^2: tTF-NGR was given as 1-hour infusion via central venous access once daily for 5 days with a subsequent rest period of 2 weeks
Arm/Group | tTF-NGR Dose: 1,0 mg/m^2 | tTF-NGR Dose: 1,5 mg/m^2 | tTF-NGR Dose: 2,0 mg/m^2 | tTF-NGR Dose: 2,5 mg/m^2 | tTF-NGR Dose: 3,0 mg/m^2 | tTF-NGR Dose: 4,0 mg/m^2 | tTF-NGR Dose: 5,0 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/2 | 0/2 | 0/8 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/2 | 2/2 | 4/8 | 4/5 | 2/3
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 2/2 | 2/2 | 6/8 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tTF-NGR Dose: 1,0 mg/m^2 (N=1) | tTF-NGR Dose: 1,5 mg/m^2 (N=2) | tTF-NGR Dose: 2,0 mg/m^2 (N=2) | tTF-NGR Dose: 2,5 mg/m^2 (N=2) | tTF-NGR Dose: 3,0 mg/m^2 (N=8) | tTF-NGR Dose: 4,0 mg/m^2 (N=5) | tTF-NGR Dose: 5,0 mg/m^2 (N=3)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) — Troponin T hs increased (grade 3, according to CTCAE 4.0) without any clinical sequelae. The increase was reversible. Troponin T hs increase was related to tTF-NGR and defined DLT.
Transient ischaemic attack (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One patient developed a reversible TIA upon treatment, which was of grade 2 according to CTCAE 4.0
Deep vein thrombosis (DVT) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 patient developed a DVT in the brachiocephalic, the jugular, and the subclavian vein. This was possibly related to tTF-NGR, but also catheter-related, 1 patient developed a grade 2 DVT in the leg, which was related to tTF-NGR. Both were reversible.
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — not drug related
Ataxia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not drug related
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — not drug related
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — tumor pain; not drug related
Lower gastrointestinal haemorrage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — not drug related
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not drug related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tTF-NGR Dose: 1,0 mg/m^2 (N=1) | tTF-NGR Dose: 1,5 mg/m^2 (N=2) | tTF-NGR Dose: 2,0 mg/m^2 (N=2) | tTF-NGR Dose: 2,5 mg/m^2 (N=2) | tTF-NGR Dose: 3,0 mg/m^2 (N=8) | tTF-NGR Dose: 4,0 mg/m^2 (N=5) | tTF-NGR Dose: 5,0 mg/m^2 (N=3)
Haemoptysis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha 1 foetoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholinesterase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasmin inhibitor decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Antithrombin III decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — stands for Troponin T hs, which was actually measured
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
International normalized ratio increased (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acitvated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection: Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02902237/Prot_SAP_000.pdf